CLINICAL TRIAL: NCT01325740
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose of STX107 in Adults With Fragile X Syndrome
Brief Title: A Study to Assess the Tolerability of a Single Dose of STX107 in Adults With Fragile X Syndrome
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: pending further evaluation
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107FX201
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- STX107 10 mg (Active Comparator)
  Interventions: Drug: STX107
- Placebo (Placebo Comparator)
  Interventions: Drug: STX107
- STX107 30 mg (Active Comparator)
  Interventions: Drug: STX107

INTERVENTIONS:
Drug: STX107 — STX107 10 mg single dose po capsule, STX107 30 mg single dose po capsule, Placebo single po capsule

SUMMARY:
The study will consist of a Screening period (up to 14 days), a Treatment period, and a Follow-Up period. Sixteen subjects will be enrolled into two sequential dose cohorts - 10 or 30 mg (or matching placebo) across four study centers.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 18 to 50 years of age, inclusive.
* Molecular documentation of the full fragile X mutation.

Exclusion Criteria:

* Subjects with a history of seizure disorder who are, in the opinion of the Investigator and Medical Monitor, not currently considered to be well controlled.
* Subjects currently being treated with psychoactive medications (including stimulants and anxiolytics).
* Subjects with any condition, including alcohol and drug abuse, which might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. 4. Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Subjects who, in the Investigator's opinion, might not be suitable for the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events will be monitored for tolerability | 1 day
  physical exam, laboratories, collection of adverse events

SECONDARY OUTCOMES:
Blood levels of STX107 will be measured to define pharmacokinetics | 1 day

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - University of California-Davis, M.I.N.D. Institute, Sacramento, California
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - Emory University School of Medicine, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois